CLINICAL TRIAL: NCT06093165
Title: RE-irradiation of Diffuse MIdline Glioma paTients
Acronym: REMIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); Radiumhospitalet, Oslo University Hospital (Unknown)
Responsible Party: Principal Investigator, Maja Maraldo, Consultant, Head of breast and paediatric radiotherapy, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMIT
Record Dates: First submitted 2023-09-08; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Diffuse Midline Glioma, H3 K27M-Mutant; Diffuse Intrinsic Pontine Glioma; Diffuse Glioma; Pontine Tumors; Thalamic Tumor; Brain Tumor, Pediatric
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Brain Stem Neoplasms; Brain Neoplasms | interventions — Re-Irradiation

STUDY DESIGN:
Masking Description: Primary radiotherapy treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Other): Primary radiotherapy 54Gy/30 fractions
  Interventions: Radiation: Re-irradiation
- B (Other): Any other dose and fractionation for primary radiotherapy than 54gy/30 fractions.
  Interventions: Radiation: Re-irradiation

INTERVENTIONS:
Radiation: Re-irradiation — 20Gy on 10 fractions

SUMMARY:
The REMIT (RE-irradiation of diffuse MIdline glioma paTients) study evaluates safety and the palliative efficacy of re-irradiation of patients with diffuse midline glioma (DMG). The study will introduce a standard re-irradiation treatment schedule for DMG patients who have progressed following primary treatment.

DETAILED DESCRIPTION:
REMIT is a non-randomized, prospective, investigator-initiated, phase II, multi-centre observational study with two inclusion groups, arm A and B. Arm A and B will be offered the same treatment.

Patients treated with primary radiotherapy 54Gy/30 fractions, either enrolled in the BIOMEDE 2.0 protocol or not, will be included in Arm A. DMG patients treated with any other total dose and fractionation than 54Gy/30F will be included in Arm B. The re-RT and follow up will be the same in both arms.

As treatment 20Gy/10 fractions is given as first time re-irradiation with extended follow up on toxicity, performance status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse midline glioma diagnosis: verified radiologically or histologically Biopsy is not mandatory for REMIT
* Age ≥ 12 months to ≤21 years.
* Min. 180 days/6 months have elapsed from the first day of the 1st RT course
* 1st course of radiotherapy
* Full recovery from all acute and subacute toxicities of 1st RT course
* Clinical progression of symptoms and/or radiographic progression
* Karnofsky performance status scale or Lansky Play Scale > 50% The performance status should not take the neurological deficits per se into account.

NB: Children and adults with a worsening performance status due to glioma-related motor deficit can be included.

* Life expectancy > 12 weeks after start of reRT
* Signed informed consent by patient and/or parents or legal guardian

Exclusion Criteria:

* Presence of leptomeningeal spread or multifocal disease on MRI at progression
* Other co-morbidity that according to the treating physician would impair participation in the study
* >1 course of radiotherapy
* Neurofibromatosis type 1
* Inability to complete the medical follow-up (geographic, social, or mental reasons)

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of re-irradiation (reRT) | 4 weeks after end of re-irradiation
  The primary endpoint will be the cumulative incidence of grade ≥4 CTCAE (The NCI Common Terminology Criteria for Adverse Events) events measured 4 weeks after the last day of reRT.

SECONDARY OUTCOMES:
The key secondary objective is to prospectively validate the palliative efficacy of reRT of DMG. Palliative efficacy is evaluated by two endpoints: overall survival and symptom relief. | 4 weeks after end of re-irradiation
  Palliative efficacy measured as overall survival will be reported as 1) from date of diagnosis to date of death by any cause, and 2) from date of first radiological and/or clinical progression to date of death by any cause.
Palliative efficacy measured as symptom relief | 4 weeks after end of re-irradiation
  Symptom relief measured by 1) clinical performance status (Karnofsky or Lansky) assessed every second week, 2) a modified PEDI score before, during and 4 weeks after reRT, 3) steroid dose levels measured every second week, and 4) quality of life monitored before, during and 4 weeks after re-irradiation with PedsQL Cancer module questionnaire.
Other secondary outcomes | through study completion
  Other secondary objectives are further defined as:
  * Image-guided characterization of the anatomical site of progression compared to the primary lesion.
  * Assessment of cumulated radiation dose to critical structures in the brain following the initial and reRT treatment.

OTHER OUTCOMES:
Exploratory analyses | through study completion
  * Delineation study A comparison of variations in delineation in tumour volume among the participating institutions. This will improve the delineation-related uncertainty and, consequently, the applied margins (and hence irradiated volume) can be diminished. This will ensure a more uniform treatment across countries.
  * The impact of reRT on the patients and their families An analysis of the value of reRT in terms of the practical, emotional, and existential impact on patients and their families. This will be done by using a qualitative method including interviewing the parents of a subgroup of the included patients.
  * Referral patterns A characterisation of referral patterns of DMG patients to reRT. This will be assessed through a screenings log of all DMG patients in the participating institutions. Date of diagnosis, date of death, reRT offered yes/no, and reason for not giving reRT will be registered prospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Maja V Maraldo, Principal Investigator — Department of oncology and radiotherapy, Copenhagen University Hospital Rigshospitalet

IPD SHARING:
Plan to Share IPD: No
All data will be collected in a RedCap database.

REFERENCES:
- [Derived] Ostergaard DE, Embring A, Sehested A, Magelssen H, Vogelius IR, Kjaersgaard M, Nysom K, Mathiasen R, Lukacova S, Maraldo MV. REMIT: Reirradiation of Diffuse Midline Glioma Patients -A Nordic Society of Paediatric Haematology and Oncology Feasibility Study. Clin Oncol (R Coll Radiol). 2025 Jan;37:103682. doi: 10.1016/j.clon.2024.103682. Epub 2024 Nov 6. PMID 39626445